CLINICAL TRIAL: NCT05267158
Title: The Cohort for Patient-reported Outcomes, Imaging and Trial Inclusion in Metastatic BRAin Disease (COIMBRA)
Acronym: COIMBRA
Status: Recruiting | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Joost J.C. Verhoeff, Principal Investigator, Radiation Oncologist, UMC Utrecht
Other Study IDs: NL67206.041.18
Record Dates: First submitted 2021-09-17; First posted 2022-03-04 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-08

CONDITIONS: Brain Metastases, Adult; Brain Neoplasms, Adult, Malignant
Keywords: radiotherapy (RT); QoL,Quality of life; Neurocognition; Brain metastases; Cranial irradiation; Neoplasm metastasis; Prognosis; Survival; Prospective
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of brain metastases is expected to increase because of better treatments of primary tumours. Novel diagnostic and therapeutic techniques are continuously being developed, all of which need thorough evaluation before they can be implemented in clinical routine. Randomized Controlled Trials are the gold standard to do so, but they have shown many challenges, especially when applied in a cancer setting.

.The 'cohort multiple Randomized Controlled Trial (cmRCT)' design is a promising design for multiple (simultaneous) randomized evaluations of experimental interventions, with potential for increased recruitment, comparability and long-term outcomes as a standard. This design will speed up the process of translating treatment innovations to the daily clinic.

DETAILED DESCRIPTION:
The COIMBRA cohort is a prospective cohort, which will serve as a facility for efficient, systematic and simultaneous evaluation of new interventions and MRI sequences and prospective outcome studies (including prediction modelling).

COIMBRA patients will be followed prospectively and information on survival, symptoms, QoL (patient and caregiver), cognition, toxicity and daily functioning in relation to treatment will be collected prospectively.

Patients will receive the regular optimal clinical care according to the current guidelines when not participating in cmRCT's.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Either radiographic and/or histologic proof of metastatic brain disease, or eligible for prophylactic cranial irradiation;
* Referred to the Department of Radiotherapy for cranial irradiation.

Exclusion Criteria:

* Mental disorder or cognitive dysfunction that hinder the patient's ability to understand the informed consent procedure and/or study details;
* Patients with severe psychiatric disorders;
* Inability to understand the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who are referred to the Department of Radiotherapy for treatment of brain metastases or for prophylactic cranial irradiation (PCI) will be asked to participate in this cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Survival | Through study completion, an average of 1 year
  Survival of participating patients will be recorded using the follow up questionnaires (returned by family members) or are derived from the Municipal Personal Records Database (in Dutch: Basisregistratie Personen (BRP))
Time and Type of re-intervention | Through study completion, an average of 1 year
  Re-intervention (re-irradiation, surgery, other); Development of neurological symptoms; Development of new metastases.
Change in toxicity after radiotherapy | Through study completion, an average of 1 year
  The toxicity will be reported by using the serious adverse event (SAE) questionnaire, every 6 months
Technical and treatment data | Through study completion, an average of 1 year
  Dose, fractions and technique of radiotherapy. All other planned and/or received treatment for brain metastases and primary tumour (i.e. systemic therapy, surgery, radiotherapy), and the characteristics there of (type, dose, duration, awake surgery, extent of surgery, complications)
  - Use of epileptic drugs, including type and dose

SECONDARY OUTCOMES:
Change in patient reported outcomes; general quality of life | Through study completion, an average of 1 year
  General quality of life will be reported by the questionnaires named C30 and EQ-5D. The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) is the instrument most frequently used to measure quality of life in cancer patients, whereas the EQ-5D is widely used to measure and evaluate general health status.
  Baseline, at 1 month, 3 months, and every subsequent 3 months, after initial radiotherapy is completed. Both the total score of the questionnaires and the individual questions are used in which we look at the difference between the measurement moments.
Change in patient reported outcomes; cancer related fatigue | Through study completion, an average of 1 year
  Cancer related fatigue is measured by using the MFI-20 questionnaire. The MFI-20 is a 20-item self-report instrument designed to measure fatigue. It covers the following dimensions: general fatigue, physical fatigue, reduced activity, reduced motivation and mental fatigue. The instrument was used in a Dutch and Scottish sample of cancer patients receiving radiotherapy
  Baseline, at 1 month, 3 months, and every subsequent 3 months, after initial radiotherapy is completed. Both the total score of the questionnaires and the individual questions are used in which we look at the difference between the measurement moments.
Change in patient reported outcomes; depression and anxiety | Through study completion, an average of 1 year
  Cancer related depression and anxiety is reported by the HADS. The Hospital Anxiety and Depression Scale (HADS) is a self-assessment questionnaire that has been found to be a reliable instrument for detecting states of anxiety and depression in the setting of hospital outpatient clinic. The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
  Baseline, at 1 month, 3 months, and every subsequent 3 months, after initial radiotherapy is completed. Both the total score of the questionnaire and the individual questions are used in which we look at the difference between the measurement moments.
Change in patient reported outcomes; disease-specific symptoms of brain metastases and (adverse) effects of their treatment | Through study completion, an average of 1 year
  Disease-specific symptoms of brain metastases and (adverse) effects of their treatment are measured by a combination of questionnaires: BN20 and CFQ. The BN20 scoring transforms 20 questions into 11 scales to assess neurological deficits (visual disorder, motor dysfunction, communication deficit), future uncertainty, and disease- and treatment-related symptoms.
  The Cognitive Failures Questionnaire (CFQ) is used in ergonomics research to measure behavioural problems associated with attentiveness and memory in everyday life.
  Baseline, at 1 month, 3 months, and every subsequent 3 months, after initial radiotherapy is completed.Both the total scores of each neurological deficit and cognitive failure and the individual questions are used in which we look at the difference between the measurement moments.
Change in caregiver reported outcomes: general quality of life | Through study completion, an average of 1 year
  General quality of life will be reported by the questionnaire EQ-5D. The EQ-5D is widely used to measure and evaluate general health status.
  Baseline, at 1 month, 3 months, and every subsequent 3 months, after initial radiotherapy of the patient is completed. Both the total score of the questionnaire and the individual questions are used in which we look at the difference between the measurement moments.
Change in caregiver reported outcomes: depression and anxiety | Through study completion, an average of 1 year
  Depression and anxiety is reported by the HADS. The Hospital Anxiety and Depression Scale (HADS) is a self-assessment questionnaire that has been found to be a reliable instrument for detecting states of anxiety and depression in the setting of hospital outpatient clinic. The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
  Baseline, at 1 month, 3 months, and every subsequent 3 months, after initial radiotherapy of the patient is completed. Both the total score of the questionnaire and the individual questions are used in which we look at the difference between the measurement moments.
Change in the caregiver burden | Through study completion, an average of 1 year
  The Caregiver Strain Index (CSI) is a tool that can be used to quickly identify families with potential caregiving concerns. It is a 13-question tool that measures strain related to care provision. There is at least one item for each of the following major domains: Employment, Financial, Physical, Social and Time. Positive responses to seven or more items on the index indicate a greater level of strain. This instrument can be used to assess individuals of any age who have assumed the role of caregiver for an older adult.
  Baseline, at 1 month, 3 months, and every subsequent 3 months, after initial radiotherapy of the patient is completed. Both the total score of the questionnaire and the individual questions are used in which we look at the difference between the measurement moments.
Patients coping and personality | Baseline
  Patients are asked to fill out the Utrechtse Coping Lijst (UCL) and the NEO Five-Factor Inventory (NEO-FFI)
Caregiver coping and personality | Baseline
  Caregivers are asked to fill out the Utrechtse Coping Lijst (UCL) and the NEO Five-Factor Inventory (NEO-FFI)
Neurocognitive functioning | We are testing this twice: once before radiotherapy and 3 months after radiotherapy
  The neuro cognitive assessment (NCA) tests that focus on the specific cognitive domains that are most sensitive to the effects of brain irradiation are used for measuring the neurocognitive functioning.
  The following domains are tested: general cognitive functioning, memory, language, executive functioning, attention, psychomotor speed, fine motor coordination, visuoconstruction, visuoperception, and social cognition. The test battery takes a maximum of 90 minutes to administer and is based upon international standards

CONTACTS AND LOCATIONS:
Overall Officials: Joost JC Verhoeff, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Coimbra Cohort (in Dutch) — http://coimbra-cohort.nl